CLINICAL TRIAL: NCT02461836
Title: An Open-Labeled, Randomized Phase II Trial of Adjuvant Chemotherapy in Combination With Stereotactic Body Radiation Therapy (SBRT) Versus Adjuvant Chemotherapy Alone for Patients After Radical Resection of Pancreatic Cancer With Advanced Stages (T3 or N1)
Brief Title: Study of Stereotactic Body Radiation Therapy for Patients After Radical Resection of Pancreatic Cancer With Advanced Stages (T3 or N1)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Principal Investigator, Liang Tingbo, Chairman of Department of Hepatobiliary & Pancreatic Surgery, Vice president of the Second Affiliated Hospital, Zhejiang University School of Medicine, Second Affiliated Hospital, School of Medicine, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YAN2015-030
Record Dates: First submitted 2015-05-28; First posted 2015-06-03 (Estimated); Last update posted 2017-04-05 (Actual); Status verified 2017-04

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Radio

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Chemo (Experimental): adjuvant chemotherapy using Gemcitabine for 6 rounds
  Interventions: Drug: Gemcitabine
- Chemo+SBRT (Experimental): SBRT is delivered prior to adjuvant chemotherapy with Gemcitabine for 6 rounds
  Interventions: Drug: Gemcitabine; Radiation: SBRT

INTERVENTIONS:
Drug: Gemcitabine — Protocol: Gemcitabine 1000mg/m2.body surface area (BSA), IV infusion for at least 30 mins, administered at Day1, Day8, Day15)
  Other Names: GEM
Radiation: SBRT — Protocol: 5 Gy/d, for 5 consecutive days
  Other Names: Radio
  Arms: Chemo+SBRT

SUMMARY:
Pancreatic cancer is one of the deadliest tumor types of the alimentary system. Resection is the only curable method to treat pancreatic cancer. However, even if radical resection is achieved, the 5-year survival rate is still low because of tumor recurrence. It's reported adjuvant radiation can prolong survival and improve quality of life after surgery. For R0 (microscopic negative margin) resection patients with advanced stages (T3 or N1), the value of adjuvant radiation is still in debate. It's warranted to explore the role of adjuvant radiation for patients after radical resection of pancreatic cancer with advanced stages (T3 or N1) in large, prospective, and randomized cohorts.

The application of Stereotactic Body Radiation Therapy (SBRT) makes radiation less harmful and more flexible. It is hoped that adjuvant SBRT may benefit post-operative patients with advanced stages and one day adjuvant SBRT combined with chemotherapy become the standard of care for pancreatic cancer patients.

DETAILED DESCRIPTION:
Pancreatic cancer is one of the deadliest tumor types of the alimentary system. Despite of the dramatic progress of diagnostic methods and surgical technics, the overall 5-year survival is still around 5%. Resection is the only curable method to treat pancreatic cancer, although only a small proportion of patients are eligible for operation. However, even if radical resection is achieved, the 5-year survival rate is only 15-20%. The main cause of death is tumor recurrence, which is as high as 50-70% in 3 years after operation. By now, it is widely accepted that pancreatic cancer is a systemic disease. Systemic treatments are recommended in neoadjuvant and adjuvant manners. It's reported adjuvant radiation can prolong survival and improve quality of life after surgery, especially for patients who undergo a R1 (microscopic positive margin) and R2 (macroscopic positive margin) resection. For R0 (microscopic negative margin) resection patients with advanced stages (T3 or N1), the value of adjuvant radiation is still in debate. Some argues adjuvant radiation after radical resection makes no effect on preventing local recurrence and metastasis but may impair patients' quality of life and overall survival. On the contrary, some other researchers draw the conclusion that adjuvant radiation may facilitate the local control of tumor recurrence in small cohorts. It's warranted to explore the role of adjuvant radiation for patients after radical resection of pancreatic cancer with advanced stages (T3 or N1) in large, prospective, and randomized cohorts.

Traditionally, radiation may take more than one month to deliver and the dosage is restricted to prevent damage to surrounding tissues. The size effects and duration impair patients' compliance. Recently, the application of Stereotactic Body Radiation Therapy (SBRT) makes radiation less harmful and more flexible. The advantages of SBRT are higher dosage of radiation, less damage to surrounding organs, and significant reduce of duration. To our knowledge, there is no big randomized clinical trial to evaluate the value of SBRT for patients after radical resection of pancreatic cancer with advanced stages (T3 or N1). It is hoped that adjuvant SBRT may benefit post-operative patients with advanced stages and one day adjuvant SBRT combined with chemotherapy become the standard of care for pancreatic cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. Male/Female subjects, age ≥ 18 years and ≤ 75 years old at the time informed consent is signed
2. Pathologically confirmed pancreatic adenocarcinoma or mixed-type pancreatic carcinoma (adenocarcinoma predominantly)
3. The operation must be radical resection (R0), with all margins negative.
4. Eastern Cooperative Oncology Group (ECOG) score: 0-2
5. Without large volume ascites or pleural effusion
6. Lab tests:

   a Complete blood cell count: HGB≥100g/L, WBC≥4×109/L, PLT≥100×109/L b Liver function: Total bilirubin≤3 x upper limit of normal range (ULN) with direct bilirubin within normal range, alanine aminotransferase (ALT) / aspartate aminotransferase (AST)≤3 c Renal function: Creatine≤1.5 x ULN or creatine clearance≥60 ml/min
7. Heart and lung function well (Eject function>55%)
8. Females of child-bearing potential must demonstrate a negative serum pregnancy test result at screening confirmed by local negative urine pregnancy dipstick within 72 hours prior to the first dose of Gemcitabine.
9. At least 30 days from major surgery before randomization, with full recovery
10. Understand and voluntarily sign an informed consent document prior to any study related assessments/procedures are conducted
11. Able to adhere to the study visit schedule and other protocol requirements

Exclusion Criteria:

1. Margin positive resections (R1 or R2)
2. Resection of recurrence pancreatic cancer
3. Other types of pancreatic cancer (non-adenocarcinoma)
4. Subjects with severe complications, can't tolerate chemotherapy in 4-12 weeks after surgery
5. Subjects with severe bone marrow suppression
6. Subjects with a history of severe lung diseases (interstitial lung disease, sarcoidosis, silicosis, idiopathic pulmonary fibrosis, pulmonary hypersensitivity pneumonitis), severe liver diseases (active hepatitis, liver cirrhosis), renal dysfunction, uncontrolled diabetes and hypertension, or multiple and severe allergies which may lead to serious complications
7. Subjects with severe heart diseases (congested heart failure, systematic coronary disease, uncontrolled arrhythmia, or myocardial infarction in 6 months)
8. Under treatment with steroids for a long time
9. Subjects with early recurrence of pancreatic cancer before initiation of chemotherapy
10. Subjects with diarrhea and infection (body temperature >38.5℃)
11. Subjects who was enrolled into another clinical study or finished another clinical study within the previous 4 weeks prior to randomization
12. Pregnant or nursing women
13. Subjects with other type of malignancies, except of curated basal cell carcinoma and carcinoma in situ of cervix which finished treatments more than half one year ago
14. Subjects having any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent them from participating in the study
15. Any condition that confounds interpreting data from the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 513 (Estimated)
Dates: Start 2015-08; Primary Completion 2020-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
disease-free survival (DFS) | Up to approximately 36 months

SECONDARY OUTCOMES:
overall survival (OS) | Up to approximately 60 months
quality of life (QOL) as assessed by the EORTC (European Organisation for Research and Treatment of Cancer) QLQ-PAN26 score | Up to approximately 60 months
safety as assessed according to NCI-CTCAE (Common Toxicity Criteria for Adverse Effects) Ver. 4 | Up to approximately 8 months
  according to NCI-CTCAE (Common Toxicity Criteria for Adverse Effects) Ver. 4

CONTACTS AND LOCATIONS:
Overall Officials: Xueli Bai, MD PHD, Principal Investigator — Zhejiang University
Locations (1):
- the second affiliated hospital of Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ma T, Bai X, Wei Q, Shui Y, Lao M, Chen W, Huang B, Que R, Gao S, Zhang Y, Chen W, Wang J, Liang T. Adjuvant therapy with gemcitabine and stereotactic body radiation therapy versus gemcitabine alone for resected stage II pancreatic cancer: a prospective, randomized, open-label, single center trial. BMC Cancer. 2022 Aug 8;22(1):865. doi: 10.1186/s12885-022-09974-7. PMID 35941566